CLINICAL TRIAL: NCT02343133
Title: A Phase 2 Single-Dose, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of HemaMax™ (rHuIL-12) in Healthy Subjects
Brief Title: Safety Study of HemaMax™ (rHuIL-12) to Treat Acute Radiation Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neumedicines Inc. (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-003; #HHSO100201100037C (Other Grant/Funding Number: BARDA)
Record Dates: First submitted 2015-01-13; First posted 2015-01-21 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Hematopoietic Syndrome Due to Acute Radiation Syndrome
Keywords: HemaMax, NM-IL-12, HSARS, Safety
MeSH Terms: interventions — Interleukin-12 Subunit p35

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HemaMax (Experimental): Single subcutaneous 12 microgram dose of HemaMax
  Interventions: Biological: HemaMax
- Placebo (Placebo Comparator): Single subcutaneous dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: HemaMax
  Other Names: rHuIL-12, NM-IL-12
  Arms: HemaMax
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether HemaMax is safe and well tolerated to support efficacy under FDA's Animal Rule to reduce the morbidity and mortality associated with the hematopoietic syndrome of acute radiation syndrome.

DETAILED DESCRIPTION:
This is a phase 2 single dose, randomized, double-blind, placebo-controlled, multi center study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of HemaMax™ (rHuIL-12) in healthy adult male and female subjects considered representative of U.S. population.

ELIGIBILITY:
Inclusion Criteria:

Male and Female healthy subjects who have signed the informed consent form must meet all of the following criteria

* ≥18 to ≤75 years of age
* Body mass index (BMI) ≥ 18 and ≤ 35 kg/m2
* Normal ECG, vital signs and laboratory test results
* Use of effective birth control method and abstinence from sex
* Negative pregnancy test and drug screen

Exclusion Criteria:

Subjects with any of the following characteristics will be considered ineligible:

* History of clinically significant renal, hepatic pulmonary, cardiovascular, cerebrovascular, gastrointestinal, metabolic, hematological, endocrine, urological, immunological, neurologic or psychiatric disorders or connective tissue disease
* Positive for human immunodeficiency virus (HIV), Hepatitis B, or surface antigen (HBsAg) or Hepatitis C antibody, tuberculosis (TB)
* Drug or alcohol addiction
* History of clinically significant allergy of any kind
* Prior use of IL-12 or HemaMax
* Use of any approved or investigational biologic agents or vaccinations of any kind in last 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of HemaMax (Number of subjects with adverse events as a measure of safety and tolerability) | 3 months
  Number of subjects with adverse events as a measure of safety and tolerability

SECONDARY OUTCOMES:
Pharmacokinetics of HemaMax (AUC, Cmax and Tmax) | 3 months
  PK parameters such as AUC, Cmax and Tmax as measures of pharmacokinetic exposure
Pharmacodynamics of HemaMax (IFN-g and CXCL-10 induction as a measure of pharmacodynamic response) | 3 months
  IFN-g and CXCL-10 induction as a measure of pharmacodynamic response
Immunogenicity of HemaMax (Anti-drug antibodies as a measure of immunogenicity) | 3 months
  Anti-drug antibodies as a measure of immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Siebers, MD, Principal Investigator — Covance Clinical Research
Locations (4):
- United States (4):
  - Covance Clinical Research Unit, Daytona Beach, Florida
  - Covance Clinical Research Unit, Evansville, Indiana
  - Covance Clinical Research Unit, Dallas, Texas
  - Covance Clinical Research Unit, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gokhale MS, Vainstein V, Tom J, Thomas S, Lawrence CE, Gluzman-Poltorak Z, Siebers N, Basile LA. Single low-dose rHuIL-12 safely triggers multilineage hematopoietic and immune-mediated effects. Exp Hematol Oncol. 2014 Apr 11;3(1):11. doi: 10.1186/2162-3619-3-11. PMID 24725395
- [Background] Gluzman-Poltorak Z, Vainstein V, Basile LA. Recombinant interleukin-12, but not granulocyte-colony stimulating factor, improves survival in lethally irradiated nonhuman primates in the absence of supportive care: evidence for the development of a frontline radiation medical countermeasure. Am J Hematol. 2014 Sep;89(9):868-73. doi: 10.1002/ajh.23770. Epub 2014 Jun 19. PMID 24852354
- [Background] Gluzman-Poltorak Z, Vainstein V, Basile LA. Association of Hematological Nadirs and Survival in a Nonhuman Primate Model of Hematopoietic Syndrome of Acute Radiation Syndrome. Radiat Res. 2015 Aug;184(2):226-30. doi: 10.1667/rr13962.1. Epub 2015 Jul 24. PMID 26207689
- [Background] Gluzman-Poltorak Z, Mendonca SR, Vainstein V, Kha H, Basile LA. Randomized comparison of single dose of recombinant human IL-12 versus placebo for restoration of hematopoiesis and improved survival in rhesus monkeys exposed to lethal radiation. J Hematol Oncol. 2014 Apr 6;7:31. doi: 10.1186/1756-8722-7-31. PMID 24708888
- [Background] Basile LA, Ellefson D, Gluzman-Poltorak Z, Junes-Gill K, Mar V, Mendonca S, Miller JD, Tom J, Trinh A, Gallaher TK. HemaMax, a recombinant human interleukin-12, is a potent mitigator of acute radiation injury in mice and non-human primates. PLoS One. 2012;7(2):e30434. doi: 10.1371/journal.pone.0030434. Epub 2012 Feb 24. PMID 22383962
- See also: Single Low-dose rHuIL-12 Safely Triggers Multilineage Hematopoietic and Immune-mediated Effects. — http://www.ehoonline.org/content/3/1/11